CLINICAL TRIAL: NCT02403375
Title: Insight Kids Study: Reaching HbA1c Targets in Children and Adolescents With Type 1 Diabetes
Brief Title: Comparing Continuous Subcutaneous Insulin Infusion With Multiple Daily Injections to Reach HbA1c Targets in Children and Adolescents With Type 1 Diabetes
Acronym: Insight Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD002177
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Subcutaneous Insulin Infusion (CSII) (Experimental): Continuous Subcutaneous Insulin Infusion (CSII) in Children and Adolescents 2-17 Years of Age
  Interventions: Device: Accu-Chek Insight Pump System

INTERVENTIONS:
Device: Accu-Chek Insight Pump System — Continuous subcutaneous insulin infusion pump

SUMMARY:
This study is to compare metabolic control, treatment satisfaction, and quality of life during continuous subcutaneous insulin infusion (CSII ) therapy with a new insulin pump system with multiple daily injections (MDI) therapy. Furthermore, this study will add clinical data originating from clinical investigation in a special population, i.e. children and adolescents of ages 2 - 17 years , to the existing clinical data of the ACCU-CHEK Insight insulin pump.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents at least 24 months of age, and not more than 17 years of age at screening
* Diagnosed with type 1 diabetes
* Diagnosis of type 1 diabetes established > 6 months before study start if >5 years of age
* Indication for insulin pump therapy according to local guidelines
* Subject's most recent HbA1c is equal or above 7.0% (53.0 mmol/mol) - measured at last assessment before screening within the past 2 months prior to the Baseline Visit into the study
* Willingness to use automated bolus advice obtained from the Accu-Chek Insight diabetes therapy system during the study
* Willingness and ability to participate and comply with study procedures

Exclusion Criteria:

* Disease or condition that in the opinion of the investigator is likely to affect compliance or the ability to complete the study
* Not willing or able to start insulin pump therapy
* Not willing to self-measure blood glucose at least four times daily
* Significantly impaired awareness of hypoglycemia
* More than one hospitalization for severe hypoglycemia during the last 12 months
* History of recurrent ketoacidosis during intensive insulin therapy
* Known strong plaster incompatibility and/or allergy
* Unstable chronic disease other than diabetes (e.g. impaired hepatic function, impaired renal function, impaired cardiac function, uncontrolled vascular complications) and any other condition interfering with the study procedures, as per Investigator´s discretion.
* If on antihypertensive, thyroid, anti-depressant or lipid-lowering medication, lack of stability on the medication for the past 2 months prior to the Baseline Visit in the study
* Chronic use of steroids in adrenal suppressive doses, other immuno-modulatory medication or chemotherapy
* Prescription medications other than insulin interfering with diabetes management
* Acute illness or abnormality (e.g. impaired vision, impaired motor function, acute pain) at the time of screening interfering with study procedures, affecting compliance, or the ability to complete the study as per Investigator´s discretion
* Either pregnant or breastfeeding
* Drug dependency
* Dependency on sponsor or Investigator (e.g. co-worker or family member)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-05-17 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Children and Adolescents of Ages 2 to 17 Years Reaching an HbA1c target of <7.5% | 26 weeks
  This HbA1c target of <7.5% proportion is statistically tested against a proportion of 25%, composed of the anticipated population proportion of 15% of children and adolescents using multiple daily insulin injections plus a safety margin of 10%.

SECONDARY OUTCOMES:
Score on Insulin Pump Questionnaire | 26 weeks
Score on Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 26 weeks
Score on Pediatric Quality of Life Inventory (PedsQL) | 26 weeks
Change from Baseline in HbA1c | 26 weeks
Change from Baseline in Blood Glucose | 26 weeks
Number of Subjects, Who Report a Diabetes-Related Adverse Event (i.e., Symptomatic Hypoglycemia, Severe Hypoglycemia, Diabetic Ketoacidosis) | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cosima Rieger, Dr., Study Director — Roche Diabetes Care
Locations (9):
- Austria (3):
  - Medical University Graz, Graz
  - Universitatsklinik fur PadiatrieI, Padiatrische Diabetologie und Endokrinologie, Innsbruck
  - Medical University of Vienna-Dept of Pediatrics, Vienna
- Germany (4):
  - Kinderkrankenhaus auf der Bult, Hanover
  - Gemeinschaftspraxis für Kinder- und Jugendmedizin, Herford
  - Practice for Pediatric and Adolescent Diabetology, Münster
  - Universitatsklinikum Tubingen, Tübingen
- United Kingdom (2):
  - Birmingham Children's Hospital Foundation Trust, Birmingham
  - St. James's University Hospital, Leeds